CLINICAL TRIAL: NCT02473146
Title: Etude Exploratoire randomisée Comparant le Traitement Par Gemtuzumab Ozogamicin /Cytarabine au Traitement Standard Par Idarubicine/Cytarabinechez Les Sujets âgés de 60 à 80 Ans et présentant Une LAM et un Caryotype Non défavorable
Brief Title: Gemtuzumab Ozogamicin+Cytarabine vs Idarubicin+Cytarabine in Elderly Patients With AML.Mylofrance 4
Acronym: ALFA1401
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Ms Juliette LAMBERT, Clinical coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-001395-65
Record Dates: First submitted 2015-04-29; First posted 2015-06-16 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; untreated; 60-80 years old; favorable and intermediate karyotype
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mylotarg Arm (Experimental): After randomization patients in the experimental arm are assigned to receive chemotherapy with:
  Gemtuzumab Ozogamicin 3 mg/m2 (maximum dose: 5 mg) per IV, 60mn on Day 1 and 4 Cytarabine 200 mg/m2 per CIV over 24h on Day 1 to 7
  Interventions: Drug: Gemtuzumab ozogamicin (GO)
- Control Arm (No Intervention): After randomization patients in the control arm are assigned to receive chemotherapy with Idarubicin 12mg/m2 per IV, 30mn on Day 1,2,3 Cytarabine 200 mg/m2 per CIV over 24h on Day 1 to 7

INTERVENTIONS:
Drug: Gemtuzumab ozogamicin (GO)
  Other Names: Mylotarg
  Arms: Mylotarg Arm

SUMMARY:
Purpose : The main objective of this study is to assess the efficacy and tolerance of the addition of repeated doses of low doses (3mg/m2) of Gemtuzumab Ozogamicin (GO) in addition with standard doses of Ara-C in previously untreated patients aged 60 to 80 years with de novo acute myeloblastic leukemia (AML) and non adverse cytogenetics. The main end point for efficacy is 2 years-event free survival. The secondary efficacy endpoints are CR/Cri rates, cumulative incidence of relapse and overall survival. The secondary endpoints for safety are early death rate (before day 30 and 60), grade 3 to 5 adverse events and severe adverse events, cardiac toxicity and quality of life. Additional secondary endpoints are treatment by covariate interactions with respect to biological characteristics present at diagnosis (CD33 positivity, cytogenetic, molecular abnormalities) or after treatment (Minimal residual disease levels). This study is an exploratory study. Patients will be allocated at inclusion with a 2/1 ratio either to receive treatment with GO and cytarabine or Idarubicin and cytarabine in a 3+7 regimen similar to the "backbone" ALFA 1200 scheme used concurrently by the ALFA group as treatment of AML patients aged >60 years.

Primary objective. The primary objective is to assess the efficacy of two doses of Gemtuzumab ozogamicin (GO) during induction and one dose of GO during first consolidation in combination with Cytarabine in elderly patients with AML in the non adverse cytogenetics-risk group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a morphologically proven diagnosis AML and both the following criteria:
* Age ≥ 60 years and < 80 years.
* Not previously treated for their disease.
* With favourable or intermediate-risk cytogenetics. (Patients with urgent clinical need to begin treatment might be included before cytogenetic results, when necessary if they do not respond to Hydroxyurea. Patients might be included if the cytogenetic results are not expected in a time limit < 5 days after AML diagnosis).
* Fit to receive intensive chemotherapy
* Cardiac function determined by radionucleide or echography within normal limits.
* Signed informed consent

Exclusion Criteria:

* M3-AML
* Presence of adverse cytogenetics (according to European LeukemiaNet recommendation.) (17) defined as one of the following abnormalities: -5/5q-, -7, t(6;9), t(v;11q23) excluding t(9;11), inv(3)(q21;q26.2) or t(3;3)(q21;q26.2), complex karyotype (3+ abnormalities)
* Secondary AML following treatment with radiotherapy or chemotherapy.
* AML following previously known myeloproliferative or myelodysplastic syndrome.
* ECOG performance status (PS) 0 to 3
* Serum creatinin level > or = 2.5N; AST and ALT level > or = 2.5N; total bilirubin level > or = 2N

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
EFS (defined as the time from randomization to the date of assessment of response if CR or Cri had not been achieved, relapse or death) | 5 years
  Endoint for the primary objective of efficacy is EFS defined as the time from randomization to the date of assessment of response if CR or Cri had not been achieved, relapse or death.

SECONDARY OUTCOMES:
Composite measure for Efficacy assessed by CR/Cri rates, cumulative incidence of relapse, overall survival. | 5 years
Composite measure for safety | 5 years
  * incidence of early deaths < day 30 and day 60,
  * grade 3 to 5 adverse events and all serious adverse events during induction and consolidation treatment
  * cardiac toxicity evaluated on cardiac ejection function evaluation by echocardiography or isotopic measure.
  * Quality of life measured by questionaries' EORTC QLQ-C30 repeated at diagnosis, after induction treatment, after the two consolidations and 3 months after the end of treatment.
  End points for treatment-by-covariate interactions are
  * at diagnosis: percentage of CD33 positivity on blast cells, measured with a standardized method, cytogenetics and most relevant molecular markers (FLT3, MLL, CEBPa, NPM1, DNMT3a.,
  * after induction and end of treatment: minimal residual disease determined by WT1 and/or NPM1 transcripts levels.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette LAMBERT, MD, Principal Investigator — Versailles Hospital; Sylvie CASTAIGNE, MD, Principal Investigator — Versailles Hospital
Locations (21):
- France (21):
  - C.H.U d'Amiens - Hôpital Sud, Amiens
  - Hôpital V. Dupouy, Argenteuil
  - CH Avicenne, Bobigny
  - CHU Caen, Caen
  - HIA Percy, Clamart
  - Hopital Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CH Dunkerque, Dunkirk
  - CH Versailles, Le Chesnay
  - Hôpital Huriez, CHU de Lille, Lille
  - CHU Limoges, Limoges
  - Hôpital de la Conception, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU d'Orléans, Orléans
  - Hopital Necker, Paris
  - Hopital St Louis, Paris
  - Hôpital Saint Antoine, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - Centre H Becquerel, Rouen
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - IGR, Villejuif